CLINICAL TRIAL: NCT05237375
Title: MIDWIZE - Strengthening Midwives to Implement and Sustain Quality Improvements to Optimise Maternity Care: A Longitudinal Observational Study in Uganda
Brief Title: MIDWIZE - Strengthening Midwives
Status: Recruiting | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: The Swedish Institute (Unknown)
Responsible Party: Principal Investigator, Helena Lindgren, Professor, Karolinska Institutet
Other Study IDs: MIDWIZE
Record Dates: First submitted 2021-12-07; First posted 2022-02-14 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Midwifery
Keywords: Midwifery, Midwife Led Care, MIDWIZE

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- The MIDWIZE model: Pregnant women giving birth during at Naguru maternity ward during the intervention period
  It's only Sub/study 2 in this PhD project which is a clinical trial and which is described onwards.
  Sub-study 2 will include all women above the age of 18 with uncomplicated full-term pregnancies and births (i.e. between weeks 37 + 0 - 42 + 0) giving birth at the delivery ward during the implementation phase.
  Data will be collected during the implementation of the quality improvement components.
  Interventions: Other: The MIDWIZE model
- The MIDWIZE model - postintervention: Pregnant women giving birth at Naguru maternity ward 3 and 6 months post intervention period.
  Sub-study 2 will include all women above the age of 18 with uncomplicated full-term pregnancies and births (i.e. between weeks 37 + 0 - 42 + 0) giving birth at the delivery ward 3 and 6 months after the implementation phase.
  Data will be collected after implementing the quality improvement components. The post-measurement data will be collected on the chosen components six months after project implementation to measure if the midwife-led quality improvement project has been sustained.
- The MIDWIZE model - scaling up: The intervention will be scaled up at three additional sites and will include all women above the age of 18 with uncomplicated full-term pregnancies and births (i.e., between weeks 37 + 0 - 42 + 0) giving birth at the delivery ward during the implementation phase.

INTERVENTIONS:
Other: The MIDWIZE model — So-called "MIDWIZE ambassadors" are planned to be appointed to lead the clinical implementation of the quality improvement components.
  Initial training workshops will be held with the ambassadors on practical aspects of the chosen components and how to explain their benefits to the units' staff. Training will also be provided on how to enhance interdisciplinary teamwork and coordinate quality improvements. The workshops will be held onsite at Naguru hospital and online via the project's "MIDWIZE virtual platform". The ambassadors will themselves hold training workshops to support midwives and other healthcare providers at the clinics during the implementation of the quality improvements components. The virtual MIDWIZE platform will contain videos, posters, presentations, and other training material that the ambassadors can utilise to enhance the units' capacity and engage their colleagues.
  Groups: The MIDWIZE model

SUMMARY:
This PhD project aims to explore how midwives can take the lead in implementing and enhancing evidence-based quality improvement (QI) components within maternal and newborn health care in Uganda.

The MIDWIZE conceptual framework will be used to understand the complexity of sustainably enhancing maternal and newborn healthcare. The project will start with a multisectoral co-creation process and subsequently involve online and onsite capacity building for midwives on selected evidence-based practices and implementation strategies. The project applies a mixed-method research approach, including focus groups discussions, interviews, quantitative data on health outcomes and a tool evaluating midwives' sense of power and autonomy.

DETAILED DESCRIPTION:
Traditionally, Quality Improvement (QI) initiatives in healthcare have often centered on the implementer's viewpoint, neglecting the active involvement of staff in shaping or leading interventions, or viewing them merely as passive objects resistant to change. Previous research in QI and organizational development indicates that when individuals or teams identify and take ownership of problems, the resulting actions are more effective and sustainable, as opposed to when solutions are imposed externally. Thus, our hypothesis was that by empowering midwives to spearhead change initiatives, involving them in the co-creation of interventions to ensure relevance and ownership, and equipping them with QI leadership and practical skills, midwives would effectively enhance healthcare service quality, foster the adoption of evidence-based practices, and ultimately improve health outcomes for women and newborns.

MIDWIZE is a model based on multisectoral collaboration to enhance evidence-based practices through Midwife-Led Care (MLC) and interdisciplinary teamwork.

Focusing on midwives as the primary health care providers at all levels of a country's maternal and reproductive health care system is an elementary part of the MIDWIZE model. Utilising midwives' potential through MLC facilitates relational, safe, cost-effective, and patient-centred care.

When additional support is required, the MLC needs to be provided in an environment that successfully takes advantage of different clinical professions' competencies. Working towards shared goals and having a clear understanding of each team member's responsibilities in an interdisciplinary team are central factors for utilising human and financial resources.

At the heart of the MIDWIZE model is enhancing the use of evidence-based practices and international guidelines for maternal and newborn health care - focusing on a healthy mother, a healthy child, a positive birth experience, and respectful care. The Z in MIDWIZE stands for the importance of "Zero separation" between the mother/birthing parent/caregiver and newborn in the early postpartum period - an evidence-based practice enhancing neonatal health outcomes, breastfeeding, and the bonding between mother/birthing parent/caregiver and child.

A prerequisite to sustainably implement or enhance these elements in a country's health system is to establish multisectoral collaborations between the four sectors (i) education, (ii) regulation, (iii) associations, and (iv) civil society. Also, the broader health system and its decision- and policymakers' readiness must be considered to create a sustainable system with continuous quality improvements within the education, regulation, and associations sectors.

General objective - this PhD project aims to explore how midwives can co-create and lead QI within midwifery and how this impacts the uptake of evidence-based practises and health outcomes for women and newborns.

Sub-study 1 - Co-creating and developing the intervention and the implementation Rationale: The involvement of stakeholders in the development of complex interventions is essential to ensure that the intervention and process are relevant, acceptable, and user friendly.

Specific objective: Describe the co-creation process and explore the needs and determinants of a midwife-led quality improvement targeting evidence-based midwifery practices.

Research Question: How do multisectoral stakeholders describe ways to implement the MIDWIZE model, how can the model be adapted to the local context and what strategies for implementation should be taken? (As the remaining parts of the intervention will be co-created, the following parts are preliminary)

Sub-study 2 - Implementation and evaluating the sustainability of the implementation Rationale: This study will explore how midwives can take the lead in implementing or enhancing evidence-based practical components of maternal care. Long-term sustainability is vital in order to maximise the potential benefits of implementation. Therefore, this study will, apart from measuring the midwives' QI projects' during the implementation phase, also measure the long-term impact six months after the project has ended. Based on the co-creation, the Midwize intervention targets three evidence-based practices where a gap between evidence and practice existed: dynamic birth positioning, empowering women in decision-making about birth positions, perineal protection, and intrapartum support. Spearheaded by a team of midwives known as the "Midwize Ambassadors," this seven-month quality improvement initiative was co-developed with expert guidance in quality enhancement and practical midwifery skills. Employing Plan-Do-Study-Act (PDSA) cycles aligned with the Model for Improvement framework, the intervention adopted a train-the-trainer methodology and conducted weekly online support sessions.

Aim: To investigate the process of a midwife-led QI intervention and the uptake of evidence-based midwifery practises.

Sub-study 3 - Outcomes Aim: To investigate the outcomes of a midwife-led QI intervention targeting evidence-based midwifery practises.

Sub-study 3 - Scaling up Aim: To explore how the Midwize intervention can be scaled up at other facilities in Kampala and what the health outcomes are for women and newborns.

Methodology Study Site Naguru maternity unit in Kampala, Uganda, is a public facility with 9000 births/year.

Study design and data collection The overall study design is a longitudinal observational study. Sub-Study 1

Focus Group Discussions (FGD) and workshops will be held in three steps:

1. Clinical staff (e.g., midwives, nurses, obstetricians, and assistant nurses), stakeholders at professional associations, academia (e.g., midwife educators, researchers, and students), and decision-makers (e.g., staff at ministry of health and hospital managers) will be included (n=36, divided into six groups). Barriers and facilitators for multisectoral collaboration will be highlighted during the workshops.
2. Members of the civil society (e.g., the projects main stakeholder - the childbearing women and their relatives) will be included in order to deliver an adequate and acceptable intervention (n=36, divided into six groups).
3. Clinical staff and managers will be included to investigate the practical implementation aspects of the project and the birth unit's adherence to national policies and clinical guidelines (n=21, divided into three groups).

Sub-Study 2 Quantitative data will be collected during and after implementing the quality improvement components. The post-measurement data will be collected on the chosen components three and six months after project implementation to measure if the midwife-led quality improvement project has been sustained.

Data is collected through observations during birth and interviews with women.

Sub-study 3: Same data will be used as for Sub-study 2 Sub-study 4: Same as in sub-study 2 but at two new intervention sites and one control site.

Sample size Sub-Study 1 Part 1 - n=36 (Clinical staff, professional associations, academia, decision-makers) Part 2 - n=36 (childbearing women and their relatives) Part 3 - n=21 (clinical staff and managers) Sub-Study 2 and 3 As this is a quality improvement project, the number of participants depends on when the targeted goal is accomplished and the total number of participants can therefore not be decided on beforehand. The targeted goal for the specific unit will be decided in dialogue with staff and management.

However, a preliminary calculation with an estimated increase of the components by 25% would suggest a minimum of 266 women during the intervention and 266 women six months after the intervention to measure the long term sustainability.

Based on previous studies, the prevalence of the three components in connection with childbirth amounts to 50%. The size of the study population is based on a calculation with 80% strength and a 95% confidence interval. A clinically significant increase in the number of women giving birth with the three components of the intervention and who are satisfied with their delivery is estimated at 25%, i.e. from 50% of women to 75% of women. To achieve this level of strength, a study population of 242 women is required. With an estimated dropout rate of 10%, there will be a study population of 266 women. To study the project's long-term sustainability, a repeated measurement that includes 266 women six months after completing data collection 2 will be done.

Measurement during the implementation phase - n=266 (birthing women) Post measurement - n=266 (birthing women)

Sampling procedure Sub-Study 1 Part 1 - A targeted selection process will be applied, and people will be included based on experience, knowledge and position in the care system (i.e. decision-makers at different levels).

Part 2 - A random sampling will be made with stakeholders of the community (in this case, pregnant women or women who recently gave birth at the clinic) Part 3 - A targeted sampling with clinical staff and managers based on profession and experience

Sub-Study 2, 3 and 4 will include all women above the age of 18 with uncomplicated full-term pregnancies and births (i.e. between weeks 37 + 0 - 42 + 0).

Pre-testing No Pre-testing will be performed as this is a quality improvement project. The data collection for sub-study two will start when the implementation starts. The outcomes will be followed until sufficient data has been achieved.

Field editing of data The research midwife will fill in the data for sub-study 2, 3 and 4 in a data collection protocol, which will be entered electronically.

Missing data. The research midwife of the day will fill in any missing data in dialogue with the clinical staff. Missing data will be continuously monitored as the data sampling will be reported online (via a secured 2-step verification platform approved to share research data).

Data Management Computer packages to use. SPSS Quality control In the qualitative parts of the project, the trustworthiness of the data will be ensured by recording interviews and FGD, transcribing verbatim, triangulation by including other researchers in the team in the analysis, regular discussions on the analysis to reach a common understanding within the team.

The quantitative data quality will be checked by random control samples made by members of the research group. A statistician will be consulted during the analysis and an electronic logbook will be kept in order for external researchers to check the procedure.

Data Analysis Presentation of data The findings will be published in peer-reviewed academic journals.

Analysis Techniques Sub-Study 1 - Thematic analysis, according to Braun & Clark (2006) Sub-Study 2, 3 and 4 - SPSS will be used for descriptive and comparative analysis of the data

ELIGIBILITY:
Inclusion Criteria:

People above the age of 18 with uncomplicated singleton full-term pregnancies and births (i.e. between weeks 37 + 0 - 42 + 0).

Exclusion Criteria:

People under the age of 18, people with complications in pregnancy or with a planned c-section.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant women coming to give birth at Naguru Hospital during or after the implementation of the MIDWIZE model.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-03-10 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
The uptake of the midwives quality improvments | Through study completion, an average of 6 months and a follow up period (2 weeks) after 3 and 6months after implementation phase is completed.
  Three evidence based midiwfery practises (i) dynamic birth positions, (ii) intrapartum support and (iii) prevetion of perineal tears .
Apgar score | Through study completion, an average of 6 months and a follow up period (2 weeks) after 3 and 6months after implementation phase is completed.
  Apgar score. The Apgar score is a rapid assessment of a newborn's health, conducted one minute and five minutes after birth, evaluating their heart rate, respiratory effort, muscle tone, reflex irritability, and color. Each component is scored from 0 to 2 points, with a maximum score of 10 points.
Perineal tear | Through study completion, an average of 6 months and a follow up period (2 weeks) after 3 and 6months after implementation phase is completed.
  Perineal tear (divided in unsutured tear, sutured tear, sphinkter tear)
Episiotomy | Through study completion, an average of 6 months and a follow up period (2 weeks) after 3 and 6months after implementation phase is completed.
  Was episiotomy performed at birth
Postpartum haemorrhage | Through study completion, an average of 6 months and a follow up period (2 weeks) after 3 and 6months after implementation phase is completed.
  Postpartum haemorrhage
Neonatal and maternal deaths | Through study completion, an average of 6 months and a follow up period (2 weeks) after 3 and 6months after implementation phase is completed.
  Neonatal and maternal deaths

SECONDARY OUTCOMES:
Mothers age | Through study completion, an average of 6 months and a follow up period (2 weeks) after 3 and 6months after implementation phase is completed.
  Mothers age
Level of education | Through study completion, an average of 6 months and a follow up period (2 weeks) after 3 and 6months after implementation phase is completed.
  Level of education for mothers giving birth during the intervention.
Marital status | Through study completion, an average of 6 months and a follow up period (2 weeks) after 3 and 6months after implementation phase is completed.
  Marital status
Area of living | Through study completion, an average of 6 months and a follow up period (2 weeks) after 3 and 6months after implementation phase is completed.
  Area of living
Employment | Through study completion, an average of 6 months and a follow up period (2 weeks) after 3 and 6months after implementation phase is completed.
  Employment
Obstetric background | Through study completion, an average of 6 months and a follow up period (2 weeks) after 3 and 6months after implementation phase is completed.6months after implementation phase is completed.
  Obstetric background
Gestation week | Through study completion, an average of 6 months and a follow up period (2 weeks) after 3 and 6months after implementation phase is completed.
  Gestation week
Mode of delivery | Through study completion, an average of 6 months and a follow up period (2 weeks) after 3 and 6months after implementation phase is completed.
  Mode of delivery
Length of second stage of labour | Through study completion, an average of 6 months and a follow up period (2 weeks) after 3 and 6months after implementation phase is completed.
  Length of second stage of labour
Birth weight | Through study completion, an average of 6 months and a follow up period (2 weeks) after 3 and 6months after implementation phase is completed.
  Birth weight
Transfer to a neonatal unit | Through study completion, an average of 6 months and a follow up period (2 weeks) after 3 and 6months after implementation phase is completed.
  Transfer to a neonatal unit
Skin-to-skin care | Through study completion, an average of 6 months and a follow up period (2 weeks) after 3 and 6months after implementation phase is completed.
  the number of minutes of skin-to-skin observed and documented by a Research Assisatant. Maximum observation time is 1hour.

CONTACTS AND LOCATIONS:
Overall Officials: Helena Lindgren, PhD, Principal Investigator — Karolinska Institutet
Locations (4):
- Uganda (4):
  - CUFH Naguru, Kampala, Naguru
  - Kawalla Hospital, Kampala
  - Kawempe Hospital, Kampala
  - Kisenye Hospital, Kampala

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berta M, Lindgren H, Christensson K, Mekonnen S, Adefris M. Effect of maternal birth positions on duration of second stage of labor: systematic review and meta-analysis. BMC Pregnancy Childbirth. 2019 Dec 4;19(1):466. doi: 10.1186/s12884-019-2620-0. PMID 31801479
- [Background] Hailemeskel S, Alemu K, Christensson K, Tesfahun E, Lindgren H. Health care providers' perceptions and experiences related to Midwife-led continuity of care-A qualitative study. PLoS One. 2021 Oct 14;16(10):e0258248. doi: 10.1371/journal.pone.0258248. eCollection 2021. PMID 34648571
- [Background] Nove A, Friberg IK, de Bernis L, McConville F, Moran AC, Najjemba M, Ten Hoope-Bender P, Tracy S, Homer CSE. Potential impact of midwives in preventing and reducing maternal and neonatal mortality and stillbirths: a Lives Saved Tool modelling study. Lancet Glob Health. 2021 Jan;9(1):e24-e32. doi: 10.1016/S2214-109X(20)30397-1. Epub 2020 Dec 1. PMID 33275948
- [Result] Blomgren J, Wells MB, Erlandsson K, Amongin D, Kabiri L, Lindgren H. Putting co-creation into practice: lessons learned from developing a midwife-led quality improvement intervention. Glob Health Action. 2023 Dec 31;16(1):2275866. doi: 10.1080/16549716.2023.2275866. Epub 2023 Nov 6. PMID 37930253
- [Derived] Blomgren J, Wells MB, Amongin D, Erlandsson K, Wanyama J, Afrifa DA, Lindgren H. Improving apgar scores and reducing perineal injuries through midwife-led quality improvements: an observational study in Uganda. BMC Public Health. 2025 Jan 3;25(1):19. doi: 10.1186/s12889-024-21137-w. PMID 39754106